CLINICAL TRIAL: NCT07395466
Title: Improving Weight Loss in Healthy Adults With Overweight and Obesity: An Artificial Intelligence-assisted Dietary Prediction and Prevention System With Continuous Glucose Monitoring
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Jocelyn Chew, Assistant Professor, National University Health System, Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NUS-IRB-2023-597
Record Dates: First submitted 2025-06-24; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Overweight , Obesity; Overweight or Obese Adults; Obesity; Overweight and/or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- eTRIP smartphone application (Experimental): Intervention group 1 involves using the eating behaviour trigger-response inhibition program(eTRIP) smartphone application for 10 weeks, where participants will need to take pictures of their food items as part of their food logging and may also engage with app-based activities to build self-regulatory skills in sticking to their weight loss plans. Additionally, participants will also apply a continuous glucose monitoring (CGM) sensor on their arm and taught how to scan the CGM sensor so that they can monitor their glucose levels for the first 10 days.
  Interventions: Behavioral: eTRIP
- FatSecret smartphone application (Sham Comparator): Intervention group 2 involves using the FatSecret smartphone application for participants to monitor their calorie intake, without any continuous glucose monitoring.
  Interventions: Other: FatSecret
- Control (No Intervention): Control group will not receive any smartphone application or continuous glucose monitoring.

INTERVENTIONS:
Behavioral: eTRIP — Intervention group 1 involves using the eating behaviour trigger-response inhibition program(eTRIP) smartphone application for 10 weeks, where participants will need to take pictures of their food items as part of their food logging and may also engage with app-based activities to build self-regulatory skills in sticking to their weight loss plans. Additionally, participants will also apply a continuous glucose monitoring (CGM) sensor on their arm and taught how to scan the CGM sensor so that they can monitor their glucose levels for the first 10 days.
  Arms: eTRIP smartphone application
Other: FatSecret — Intervention group 2 involves using the FatSecret smartphone application for participants to monitor their calorie intake, without any continuous glucose monitoring.
  Arms: FatSecret smartphone application

SUMMARY:
This study aims to examine the effectiveness of a novel dietary lapse prediction and prevention self-regulation app called the eating behaviour trigger-response inhibition program (eTRIP), and the addition of continuous glucose monitoring (CGM), on healthy eating and weight loss in people with overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

1. are 21-65 years old
2. have BMI ≥23 kg/m2
3. can comprehend the English language
4. uses a smartphone that can download apps
5. are willing to perform continuous glucose monitoring (CGM) using the Dexcom continuous glucose monitoring system
6. willing to travel to the National University of Singapore (NUS)
7. able to provide informed consent

Exclusion Criteria:

1. are using/intend to use other apps for weight loss;
2. are pregnant or lactating (as it would affect weight change and caloric needs)
3. are diagnosed severe mental disorders (e.g. major depressive disorder and schizophrenia)
4. are on prescribed meal replacements or pharmacotherapy
5. have serious medical conditions
6. are scheduled for any kind of surgery within the next 6 months

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Height | At weeks 0, 10 and 24.
  Taken using a wall mounted measuring tape.
Weight | At weeks 0, 10 and 24.
  Taken using InBody 120
Waist Circumference | At weeks 0, 10 and 24.
  Taken using a measuring tape.
BMI | At weeks 0, 10 and 24.
  Taken using InBody 120
Self regulation of Eating Behaviour Questionnaire (SREBQ) | At weeks 0, 10 and 24.
  The Self-Regulation of Eating Behaviour Questionnaire (SREBQ) is a validated self-administered instrument used to assess individuals' self-regulation in relation to eating behavior. It evaluates the extent to which individuals monitor, control, and regulate their eating behaviors in everyday contexts. Higher scores indicate greater self-regulation of eating behavior.

SECONDARY OUTCOMES:
Patient Health Questionnaire-2 (PHQ-2) | At weeks 0, 10 and 24.
  The Patient Health Questionnaire - 2 item (PHQ-2) is a validated self-administered screening questionnaire used to assess the frequency of depressive symptoms over the past two weeks. Higher scores indicate greater depressive symptom severity.
Euro Quality of life 5 Dimensions-5 Levels (EQ-5D-5L) | At weeks 0, 10 and 24.
  The EuroQol 5 Dimensions - 5 Levels (EQ-5D-5L) is a standardized self-administered instrument used to assess health-related quality of life. It measures five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each with five response levels.
Generalized Anxiety Disorder 2-item (GAD-2) | At weeks 0, 10 and 24.
  The Generalized Anxiety Disorder - 2 item (GAD-2) is a validated self-administered screening questionnaire used to assess the frequency of core anxiety symptoms over the past two weeks. Higher scores indicate greater anxiety symptom severity.
Percentage Body Fat | At weeks 0, 10 and 24.
  Taken using InBody 120.
Body Fat Mass | At weeks 0, 10 and 24.
  Taken using InBody 120.
Three Factor Eating Questionnaire (TFEQ) | At weeks 0, 10 and 24.
  The Three-Factor Eating Questionnaire (TFEQ) is a validated self-administered instrument used to assess eating-related behaviors. It measures three domains: cognitive restraint of eating, uncontrolled eating, and emotional eating. Higher scores indicate greater levels of the respective eating behavior.
International Physical Activity Questionnaire Short-Form (IPAQ-SF) | At weeks 0, 10 and 24.
  The International Physical Activity Questionnaire - Short Form (IPAQ-SF) is a validated self-administered questionnaire used to assess self-reported physical activity levels. It captures the frequency and duration of walking, moderate-intensity activity, and vigorous-intensity activity performed over the past 7 days.
Self-Report Behavioural Automaticity Index (SRBAI) | At weeks 0, 10 and 24.
  The Self-Report Behavioural Automaticity Index (SRBAI) is a validated self-administered questionnaire used to assess the automaticity of behavior. It evaluates the extent to which a behavior is performed automatically, with little conscious thought or deliberation. Higher scores indicate greater behavioral automaticity.
Consideration of Future Consequences Scale (CFCS-6) | At weeks 0, 10 and 24.
  The Consideration of Future Consequences Scale - 6 item (CFCS-6) is a validated self-administered questionnaire used to assess the extent to which individuals consider the potential future outcomes of their current behaviors. It evaluates the degree to which individuals weigh immediate versus future consequences when making decisions. Higher scores indicate greater consideration of future consequences.
Skeletal Muscle Mass | At weeks 0,10 and 24.
  Taken using InBody 120.
Visceral Fat Level | At weeks 0, 10 and 24.
  Taken using InBody 120.
Big Five Inventory - 44 item (BFI-44) | At weeks 0, 10 and 24.
  The Big Five Inventory - 44 item (BFI-44) is a validated self-administered questionnaire used to assess personality traits across five domains: openness, conscientiousness, extraversion, agreeableness, and neuroticism. Higher scores indicate greater expression of the respective personality traits.

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No